CLINICAL TRIAL: NCT01511094
Title: Goniocurettage as First Choice of Surgical Treatment in Chronic Open-Angle Glaucoma: Outcomes and Complications
Acronym: GC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Tiago Tomaz de Souza, Principal Investigator, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gonio-32
Record Dates: First submitted 2011-10-14; First posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Open-Angle Glaucoma; Surgery
Keywords: ab-interno trabeculectomy,; intraocular pressure,; open angle glaucoma; trabeculectomy; Goniocurettage; Non-Filtering Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eye Surgery (Experimental): Goniocurettage was used to treat open angle glaucoma patients
  Interventions: Procedure: Goniocurettage

INTERVENTIONS:
Procedure: Goniocurettage — Ab interno surgery consisting on scraped away the trabecular tissue from the angle (goniocurettage) removing segments of pathologically altered trabecular meshwork from the scleral sulcus
  Other Names: Ab interno glaucoma precedure; Open angle glacuoma surgery; Non filtering glaucoma procedure

SUMMARY:
The study has the purpose to evaluate the effectiveness and safety of the goniocurettage as a first choice of surgical treatment for primary open-angle glaucoma (POAG) in patients with good vision.

DETAILED DESCRIPTION:
A prospective study in 33 eyes (32 patients) with uncontrolled open angle glaucoma under clinical treatment. The trabecular tissue was scraped away from the angle (goniocurettage) in about 100 degrees by means of an instrument similar to a microchalazion curette. The goniocurettage was done under direct visualization of the angle through a gonioscopy lens (Swan-Jacob) and a surgical microscope. Using the 17.0 SPSS software the investigators compared the intraocular pressure, the numbers of antiglaucomatous medications, the best correct visual acuity, the development of cataract, the central corneal thickness,the impact on the visual field, the impact on the optic nerve head and the central corneal endothelial cell density before and after the goniocurettage, and the intra and post operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Disc and/or visual field findings consistent with Primary Open Angle Glaucoma
* Uncontrolled intraocular pressure (≥21 mm Hg) or progressive glaucomatous neuropathy despite maximum tolerated medical therapy
* 40 years old or over
* Visual acuity higher than 0.2
* Open angles (greater or equal to Shaffer grade II)

Exclusion Criteria:

* Previous ocular surgery
* History of glaucoma laser treatment
* History of ocular trauma
* Cyclodestructive procedures
* Corneal edema or opacities
* Endothelial decompensation
* History of uveitis
* Secondary glaucoma
* neovascularization of the iris or angle
* Congenital anterior segment abnormalities
* Anatomically confusing angles without clear definition of the scleral spur or meshwork and inability to maintain follow-up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular Pressure | Change from Baseline in Intra Ocular Pressure at 20 months
  The mean of at least three measures at 8:00 am two weeks before surgery. After intervention, the Intra Ocular Pressure was measured on the day after, one week after, two weeks after and every month at the same time until the end of the study (an expected average of 20 months).

SECONDARY OUTCOMES:
Central Corneal Thickness | Two weeks before, six months after and one year after intervention
Central corneal endothelial cell density | Two weeks before, six months after intervention and one year after intervention
Best correct visual acuity | Two weeks before, six months after and one year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tiago T Souza, MD, Principal Investigator — Federal University of Minas Gerais; Sebastiao Cronemberger, PhD, Study Director — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Jacobi PC, Dietlein TS, Krieglstein GK. Technique of goniocurettage: a potential treatment for advanced chronic open angle glaucoma. Br J Ophthalmol. 1997 Apr;81(4):302-7. doi: 10.1136/bjo.81.4.302. PMID 9215060
- [Background] Jacobi PC, Dietlein TS, Krieglstein GK. Goniocurettage for removing trabecular meshwork: clinical results of a new surgical technique in advanced chronic open-angle glaucoma. Am J Ophthalmol. 1999 May;127(5):505-10. doi: 10.1016/s0002-9394(98)00448-6. PMID 10334341
- [Background] Jacobi PC, Dietlein TS, Krieglstein GK. Microendoscopic trabecular surgery in glaucoma management. Ophthalmology. 1999 Mar;106(3):538-44. doi: 10.1016/S0161-6420(99)90113-6. PMID 10080211
- [Background] Johnson DH, Johnson M. How does nonpenetrating glaucoma surgery work? Aqueous outflow resistance and glaucoma surgery. J Glaucoma. 2001 Feb;10(1):55-67. doi: 10.1097/00061198-200102000-00011. PMID 11219641
- [Background] Minckler D, Baerveldt G, Ramirez MA, Mosaed S, Wilson R, Shaarawy T, Zack B, Dustin L, Francis B. Clinical results with the Trabectome, a novel surgical device for treatment of open-angle glaucoma. Trans Am Ophthalmol Soc. 2006;104:40-50. PMID 17471324